CLINICAL TRIAL: NCT04727346
Title: Assessment of Post-surgical Improvement in Obstructive Sleep Apnea Patients After Imaging of Upper Respiratory Airway Using Cone Beam Computed Tomography (CBCT) and Drug-Induced Sleep Endoscopy (DISE) Versus Drug-Induced Sleep Endoscopy Only: A Validity Study
Brief Title: Evaluation of Post-surgical Improvement in OSA Patients After Imaging of Upper Airway Using CBCT and DISE vs DISE Only
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marco Emad Shawky Isaac, PhD student, Cairo University
Other Study IDs: OCS05051989
Record Dates: First submitted 2021-01-17; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: CBCT, OSA, DISE
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: CBCT and DISE
  Interventions: Radiation: CBCT; Procedure: DISE
- Control Group: DISE only
  Interventions: Procedure: DISE

INTERVENTIONS:
Radiation: CBCT — Cone Beam Computed Tomography
  Groups: Study Group
Procedure: DISE — Drug Induced Sleep Endoscopy

SUMMARY:
CBCT is considered an innovative imaging modality that can view the upper respiratory airway anatomy in a 3D manner. Recent studies tried to evaluate the accuracy of CBCT in analyzing the upper respiratory airway and its related structures. Although, most of these studies aimed to evaluate the 3D imaging of upper respiratory airway in OSA patients and their healthy counterparts, the determination of its level of collapse with the aid of CBCT wasn't clearly evaluated.

DISE is considered a dynamic approach to determine the level of upper respiratory airway collapse accurately, but CBCT can offer better evaluation of anatomical upper respiratory airway characteristics and morphology which in turn affects treatment planning and patients' satisfaction after surgery. The hypothesis is agreed with other studies who found that retroglossal collapse appears more frequently during the end of expiration imaged by dynamic MRI.

Our hypothesis is the validity of CBCT in determining the level of collapse through assessing different orthogonal planes at end of inspiration and expiration especially in those patients having a tongue/palate interaction or lengthy palate where this anatomical variation wasn't been probably evaluated with DISE.

DETAILED DESCRIPTION:
In this validity two-arm study, a total (n) patients will be included; all are diagnosed with OSA and will undergo surgical treatment after appropriate planning. Patients will be classified into two equal groups with allocation ratio (1:1). Patients of the study group will be examined after scanning with CBCT at both ends of expiration and inspiration and DISE. Control group patients will be examined by DISE only. After discussing the treatment plan with the patient and educating the patient with all the data needed, an arabic consent form will be signed by the willing participants.

These (n) patients will be selected by the ENT specialist according to the following;

* A multidisciplinary approach will be performed to diagnose OSA patients who are indicated for surgery. Firstly, a comprehensive assessment of patients' history will be performed; including evaluation of all risk factors and complete sleep history.
* Epworth Sleepiness Scale (ESS) which consists of eight section questionnaire that defines the frequency of an individual to fall asleep during regular daily activities will be obtained from the patients.
* Afterward, a proper physical examination will be performed including a thorough clinical examination of the oropharynx, nasopharynx, and hypopharynx to evaluate any anatomical abnormalities as impotency of the nasal airway, elongated soft palate or uvula, enlarged lingual tonsils, and any other pathological conditions of tongue, palate, and tonsils.
* Then, Polysomnography (PSG) (sleep study) will be performed to allow proper evaluation of normal and abnormal physiological sleep episodes. Apnea/Hypoapnea Index (AHI) will be reported to detect the severity of OSA and patients were classified into mild (AHI = 5-14/ hour), moderate (AHI = 15-30 / hour) and severe (AHI >30 / hour).
* All patients in both groups will undergo upper airway surgery, DISE will be performed by the same ENT surgeon to detect the level of collapse in the upper airway which will be assessed by LwPTL and VOTE classifications, emphasizing on the primary structures contributing at upper airway collapse, either alone or in combination: the larynx, palate, tongue and pharyngeal lateral walls.
* Study group participants only will be scanned by CBCT twice; once at the end of inspiration and the other at the end of expiration while they are gently holding their breath for as long as possible.
* In the study group, surgical procedures decision will be taken after appropriate assessment to sites of collapse in CBCT views at both ends of expiration and inspiration vies in combination to DISE.
* Finally, strict post-operative instructions will be given to patients of both group and a 3 months follow up would be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age is more than 18 years old.
* Patients are indicated for upper respiratory airway surgery based on adequate history taking, proper clinical examination, and sleep study.
* Patients refusing Continuous Positive Airway Pressure (CPAP) treatment.
* Systemically medically free patients.

Exclusion Criteria:

* Patients who are refusing the surgical approach as a treatment plan option.
* Patients who have undergone previous surgeries in the upper respiratory airway.
* Pregnant women.
* Patients who didn't follow post-operative instructions.
* Patients who are not able to come for the follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstructive Sleep Apnea Patients Indicated for Surgery
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-05-22 (Estimated); Study Completion 2022-07-22 (Estimated)

PRIMARY OUTCOMES:
Post-surgical improvement | 3 months after the surgery
  through Mean Apnea/Hypoapnea Index (AHI) reduction percentage by Polysomnography (PSG) (sleep study)

SECONDARY OUTCOMES:
Level of Collapse of the upper respiratory airway | immediately after performing both DISE and CBCT
  through LwPTL Classification
The volume of the upper respiratory airway. | through study completion, an average of 1 year
  through CBCT images (Invivo5 software)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Isaac, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pang KP, Baptista PM, Olszewska E, Braverman I, Carrasco-Llatas M, Kishore S, Chandra S, Yang HC, Wang CMZ, Chan YH, Pang KA, Pang EB, Rotenberg B. Does drug-induced sleep endoscopy affect surgical outcome? A multicenter study of 326 obstructive sleep apnea patients. Laryngoscope. 2020 Feb;130(2):551-555. doi: 10.1002/lary.27987. Epub 2019 Apr 17. PMID 30993741

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT04727346/Prot_SAP_ICF_000.pdf